CLINICAL TRIAL: NCT03668067
Title: Refractive and Strabismic Amblyopia Risk Factors Detected by Infrared Photoscreener and School Bus Skiascopy
Brief Title: Performance of 2WIN Photoscreener With Corneal Reflex Compared to School Bus Retinoscopy by AAPOS Guidelines
Acronym: 2WINbus
Status: Completed | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: ABCD 2WIN bus
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Refractive Errors; Amblyopia; Strabismus; Development Delay
MeSH Terms: conditions — Refractive Errors; Amblyopia; Strabismus; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Photoscreener (2WIN): Accommodation, refraction and ocular alignment are estimated by infrared photoscreener using the photoscreener device. Photoscreener screening makes use of light crescent quantification from off-axis flash-to-lens in a camera.
  Interventions: Device: 2WIN photoscreener
- school bus skiascopy: Refractive error estimated by child-friendly skiascopy rack holding lenses from +1.00 D to +10.00 D and -5.00 D. Skiascopy is a common, old-fashioned form of retinoscopy.

INTERVENTIONS:
Device: 2WIN photoscreener — conventional infrared off-axis photoscreener
  Groups: Photoscreener (2WIN)

SUMMARY:
Pediatric eye patients receive infrared photoscreener screening and skiascopy as a part of routine examination to compare ability to detect amblyopia risk factors.

DETAILED DESCRIPTION:
Patients: Pediatric eye and adult strabismus patients undergoing routine examinations in a private ophthalmology practice.

Interventions: Infrared photoscreener / remote autorefractor such as 2 Winner (2WIN) ("Adaptica" - Padova, Italy) without and with infrared corneal reflex occluder. Child-friendly skiascopy before and after cycloplegic refraction.

Outcome: Amblyopia Risk Factors from comprehensive eye exam including refraction and strabismus.

Risk factors defined by American Association for Pediatric Ophthalmology and Strabismus (AAPOS) 2003 and 2013 guidelines.

**Please note that 2 Winner has nothing to do with actual device, but was required by the Clinical Trials Web entry.**

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing eye examination

Exclusion Criteria:

* none

Ages: 1 Week to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: male and female children and adults with strabismus developmental delay is NOT excluded
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Amblyopia Risk Factor (refractive error and/or strabismus) | 2 hours or less: Screening and Gold Standard Exam performed the same day, usually within the same hour.
  Whether pre-defined, age-related risk factor is present. AAPOS has published standard levels of these refractive errors or binocular misalignment that render a child at risk of developing sight-threatening amblyopia.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Arnold, MD, Principal Investigator — Alaska Blind Child Discovery
Locations (1):
- Alaska Children's EYE & Strabismus, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified database on-line available
Supporting Information: Study Protocol
Time Frame: late 2018
Access Criteria: public website
URL: http://www.abcd-vision.org/references/index.html

REFERENCES:
- [Background] Tsao Wu M, Armitage MD, Trujillo C, Trujillo A, Arnold LE, Tsao Wu L, Arnold RW. Portable acuity screening for any school: validation of patched HOTV with amblyopic patients and Bangerter normals. BMC Ophthalmol. 2017 Dec 4;17(1):232. doi: 10.1186/s12886-017-0624-y. PMID 29202721
- [Background] Donahue SP, Arthur B, Neely DE, Arnold RW, Silbert D, Ruben JB; POS Vision Screening Committee. Guidelines for automated preschool vision screening: a 10-year, evidence-based update. J AAPOS. 2013 Feb;17(1):4-8. doi: 10.1016/j.jaapos.2012.09.012. Epub 2013 Jan 27. PMID 23360915
- [Background] Arnold RW, Davis B, Arnold LE, Rowe KS, Davis JM. Calibration and validation of nine objective vision screeners with contact lens-induced anisometropia. J Pediatr Ophthalmol Strabismus. 2013 May-Jun;50(3):184-90. doi: 10.3928/01913913-20130402-02. Epub 2013 Apr 9. PMID 23565714
- [Background] Arnold RW, Arnold AW, Hunt-Smith TT, Grendahl RL, Winkle RK. The Positive Predictive Value of Smartphone Photoscreening in Pediatric Practices. J Pediatr Ophthalmol Strabismus. 2018 Nov 19;55(6):393-396. doi: 10.3928/01913913-20180710-01. Epub 2018 Aug 29. PMID 30160295
- [Background] Kirk S, Armitage MD, Dunn S, Arnold RW. Calibration and validation of the 2WIN photoscreener compared to the PlusoptiX S12 and the SPOT. J Pediatr Ophthalmol Strabismus. 2014 Sep-Oct;51(5):289-92. doi: 10.3928/01913913-20140701-01. Epub 2014 Jul 8. PMID 25000209
- [Background] Arnold SL, Arnold AW, Sprano JH, Arnold RW. Performance of the 2WIN Photoscreener With "CR" Strabismus Estimation in High-Risk Patients. Am J Ophthalmol. 2019 Nov;207:195-203. doi: 10.1016/j.ajo.2019.04.016. Epub 2019 May 9. PMID 31077668
- [Derived] Arnold AW, Arnold SL, Sprano JH, Arnold RW. School bus accommodation-relaxing skiascopy. Clin Ophthalmol. 2019 Oct 8;13:1841-1851. doi: 10.2147/OPTH.S219031. eCollection 2019. PMID 31631961
- Available data/document: Individual Participant Data Set — http://www.abcd-vision.org/references/2WIN%20Bus%20de-identified%209-6-18.pdf — Public de-identified ongoing